CLINICAL TRIAL: NCT01264029
Title: Efficacy of Mindful Tai Chi Intervention on Obese and Overweight Adults: A Randomized Controlled Clinical Trial
Brief Title: Efficacy of Mindful Tai Chi on Obese or Overweight Adults: A Randomized Controlled Clinical Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 110030; 11-NR-0030
Record Dates: First submitted 2010-12-18; First posted 2010-12-21 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2012-11-05

CONDITIONS: Obesity; Adult; Healthy
Keywords: Well-Being; Tai Chi; Obesity; Mindfulness; Meditation; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Mindfulness

ARMS (4):
- Group A (Experimental): Movement meditation for 2 hours
  Interventions: Behavioral: Mindful Tai Chi Intervention
- Group B (Active Comparator): Non-moving sitting meditation for 2 hours
  Interventions: Behavioral: Mindfulness Meditation
- Group C (Active Comparator): Mall Walking for 2 hours
  Interventions: Behavioral: Mall Walking
- Group D (Active Comparator): Weekly Discussion
  Interventions: Behavioral: Weekly Discussion

INTERVENTIONS:
Behavioral: Mindful Tai Chi Intervention
  Arms: Group A
Behavioral: Mindfulness Meditation
  Arms: Group B
Behavioral: Mall Walking
  Arms: Group C
Behavioral: Weekly Discussion
  Arms: Group D

SUMMARY:
Background:

* New weight-loss intervention programs are being studied to determine their effectiveness in helping overweight and obese individuals reach a healthy weight. However, these programs often have not been tested against each other, and researchers are interested in determining which interventions are most effective both immediately and over the long term in promoting and maintaining weight loss.
* Mindful Tai Chi is a combined form of the meditative martial art tai chi and the practice of mindfulness meditation. Tai chi and mindfulness meditation both have common philosophical underpinnings that address health promotion and well-being by applying the skill of non-judgmental awareness on a moment-to-moment daily basis. More research is needed on whether Mindful Tai Chi and mindfulness meditation can help improve various health factors in overweight and obese individuals.

Objectives:

- To compare the effects of Mindful Tai Chi, mindfulness meditation, walking, or a discussion group on the weight and well being of overweight and obese participants.

Eligibility:

- Healthy individuals at least 18 years of age who are either overweight or obese (body mass index between 25 and 40), have a sedentary lifestyle (have not engaged in more than 1 hour of aerobic exercise per week within the last month), and are willing to commit to a specific weight-loss intervention program.

Design:

* This study involves four visits for collecting information and 12 weeks of research study activities.
* During the first visit, participants will hear information about the study and may ask any questions. They will be screened with a medical history and physical examination, and those eligible will be assigned to one of the four study groups: Mindful Tai Chi (MTC), Mindfulness Meditation (MM), Mall Walking (MW), or Weekly Discussion (WD) group.
* For the second visit, participants will give blood and urine samples, receive an abdominal ultrasound, ride a stationary bicycle for 5 minutes, and fill out health-related questionnaires.
* For 12 weeks, participants will be involved in the following activities depending on their group:
* MTC: Class for 2 hours per week, emphasizing the meditation aspects of tai chi. Each session will include at least 20 minutes of meditation. Participants will receive written instructions and an accompanying DVD in comparable formats specifying a minimum of 30 minutes of daily home assignment. In weeks 2 and 8, participants will have a workshop for mindfulness skill application in daily activity.
* MM: Class for 2 hours per week of mindfulness meditation. Participants will receive written instructions and an accompanying DVD in comparable formats specifying a minimum of 30 minutes of daily home assignment. In weeks 2 and 8, participants will have a workshop for mindfulness skill application in daily activity.
* MW: Participants will meet at a designated mall location once a week for 2-hour walk.
* WD: Participants will meet at the National Institutes of Health for weekly weight-loss discussion.
* For the third and fourth visits, participants will receive the same procedures as those used in the second visit. These visits will occur at the end of the 12-week activity period and at a 3-month follow up visit.

DETAILED DESCRIPTION:
Objective: The objective of this protocol is to pilot test the efficacy of a Mindful Tai Chi (MTC) intervention as an integrative approach to facilitate durable weight loss and well-being among sedentary obese and overweight individuals. Numerous interventions for obesity are available but the results are temporary, with most individuals returning to or exceeding their baseline weights. Contrasting with conventional emphases on quantitative weight reduction with factual didactics, exercise and diet, this protocol will focus on enhancing individuals integrative resources utilizing mindfulness principles facilitating changes in self healthcare behaviors.

MTC is a combined form of Tai Chi and mindfulness meditation. Tai Chi and mindfulness both have common philosophical underpinnings that address health promotion and well-being. Tai Chi is a gentle moving meditation that fosters individuals body-mind-spiritual integration through specific movements. MTC is a systemic intervention with multidimensional effects on health and well-being that facilitate healthy lifestyle by applying the skill of non-judgmental awareness on a moment-to-moment daily basis. We hypothesize improvements in health and well-being variables of the participants.

Study population: Healthy ambulatory volunteers 18 years and older with BMI between 25 and < 40 will be recruited from the greater Washington area. Exclusion criteria include mental or physical health limitations that impede participation in the treatments or assessment of outcome variables.

Design: A randomized controlled clinical trial: comparing the MTC group to an active health education (HE) control group. These groups will participate in the assigned activities in a 90 minute session twice a week for 10 weeks. All groups will be assessed at baseline and upon completion of the treatments at week 10 and at a 2 month follow-up.

Outcome measures: The primary outcomes are changes in weight and multiple domains of well-being. BMI and intra-abdominal fat by abdominal ultrasound will measure weight changes. Physical well-being variables include biomarkers (lipid profile, BP, CRP, Leptin, IL 6, and A1C), aerobic fitness from VO(2) max measurement with 6 to 10 minutes of a treadmill test, and telomerase activity in leukocytes. A battery of questionnaires will measure psychological, cognitive-affective, socio-spiritual and overall well-being. Secondary outcomes include mindfulness quality and lifestyle indices.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Male or female volunteers ages 18 and older with BMI between 25.0 and < 40 and a sedentary lifestyle. Sedentary lifestyle is defined as less than 60 minutes of deliberate health activities per week within the last month.
* Willing to be assigned to one of the two arms.
* Able to understand 5th grade English
* General ability and willingness to follow directions for home assignment.
* TC and mindfulness meditation naive within the last 2 years
* Can move all extremities freely and can ambulate without assistance.
* Weight fluctuation < 10 lbs during the last month

EXCLUSION CRITERIA:

* Individuals with psychological, physical, neuro-cognitive, or muscular impairments that interfere with MTC or HE participation. A diagnosis of psychosis, affective disorder, myocardial infarction, cardiovascular accident, or hospitalization related to other serious illnesses within the last 12 months and/or by H&P examination conducted by MD or CRNP at NIH.
* Contradiction to blood drawing such as clotting disorders.
* Active drug or alcohol abuse: self report of any illicit drug or > 2 glasses of wine or equivalent alcohol consumption per day or positive urine drug test.
* Mini Mental Status Exam (MMSE) scores < 24.
* Peripheral neuropathies and neuro-musculoskeletal conditions that may increase the fall risk.
* Pregnancy as revealed by self report or positive urine test.
* Severe vertigo or Meniere s disease or history of known equilibrium problems.
* Taking weight loss medication or starting to take weight loss medicine during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-12-09; Primary Completion 2012-11-05 (Actual); Study Completion 2012-11-05 (Actual)

PRIMARY OUTCOMES:
Weight loss (BMI, Intra-abdominal fat)
Well-being (physical, psychological, cognitive-affective, social-spiritual, and overall)

SECONDARY OUTCOMES:
Mindfulness
Lifestyle indices
Telomerase activity (exploratory variable)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond A Dionne, D.D.S., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Alperson SY. Tai Chi philosophy and nursing epistemology. ANS Adv Nurs Sci. 2008 Jan-Mar;31(1):E1-E15. doi: 10.1097/01.ANS.0000311532.65941.b8. PMID 20531257
- [Background] Andersson J, Boman K, Jansson JH, Nilsson TK, Lindahl B. Effect of intensive lifestyle intervention on C-reactive protein in subjects with impaired glucose tolerance and obesity. Results from a randomized controlled trial with 5-year follow-up. Biomarkers. 2008 Nov;13(7):671-9. doi: 10.1080/13547500802661266. PMID 19096961
- [Background] Arias AJ, Steinberg K, Banga A, Trestman RL. Systematic review of the efficacy of meditation techniques as treatments for medical illness. J Altern Complement Med. 2006 Oct;12(8):817-32. doi: 10.1089/acm.2006.12.817. PMID 17034289